CLINICAL TRIAL: NCT02005913
Title: A Novel Patent Platform of Detection of Circulating Tumor Cells to Early Detect Colorectal Cancer Recurrence
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201309068RINC
Record Dates: First submitted 2013-12-04; First posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Colorectal Cancer (CRC)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The best strategy to prevent colorectal cancer (CRC) death lies in early detection and early treatment at the local disease status of tumor. After curative resection of tumor, there are about 5~10% of stage I, 20~30% of stage II and 40~50% of stage III patients suffering metastasis during subsequent follow-up periods. Although carcinoembryonic antigen (CEA) is the most widely used biomarker for postoperative monitoring of recurrence on asymptomatic patients, it is difficult to use CEA as biological marker to identify the population with high recurrent risk in patients with early-stage cancer because lower than half of patients with early-stage cancer do not have CEA elevation. For improving the survival of patients with early-stage CRC, we need effort to search more useful biological markers to predict the risk of tumor recurrence and to select out patients with high recurrent risk to receive preventive adjuvant therapy.

Circulating tumor cells (CTCs) in the blood play an essential role in cancer metastasis. Hence, the detection of CTCs and subsequent analysis can potentially revolutionize the cancer care ranging from screening, diagnosis, monitoring, to drug selection and so on. In the past decade, many methods using magnetic beads (CellSearch), filtration (RareCelletc), or flow cytometry have been developed but all of them have the shortcomings from low sensitivity, low purity, to unable to retrieve cells for downstream molecular analysis and cell culture. Recently, a biomimetic affinity based microfluidic platform has overcome abovementioned technical challenges. Importantly, by using only 2 ml of peripheral blood, Sinica's team has shown that the enumeration of CTCs increases with the CRC disease progression, where the mean CTC counts are 3, 15, 29 and 60 per ml for the stages I, II, III and IV, respectively. The results imply that monitoring CTC enumeration serially may serve as a prediction marker to identify the CRC patients with high probability of recurrence. The aims of this study are toestablishing CTC platform standard operation protocol (SOP) that leads to certification of ISO 13485 and to establish CTC criteria and evaluate its prediction power of early detection of colorectal cancer recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of colorectal cancer

Exclusion Criteria:

* age younger than 20
* Pregnancy
* Inmates

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diagnosed colorectal cancer patient
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2014-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
tumor recurrence | 1, 3, 6, 9 and 12 months post-surgery and 2 and 3 years after surgery as part of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Ting Chang, MD.PhD, Principal Investigator — Visting stuff of national taiwan university hospital; National Taiwan University NTUH, Study Chair — Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan